CLINICAL TRIAL: NCT05965687
Title: Normobaric Hyperoxia Combined With Intravenous Thrombolysis for Acute Ischemic Stroke (OPENS-3)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ji Xunming,MD,PhD (Other)
Collaborators: Beijing Friendship Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Tongren Hospital (Other); People's Hospital of Beijing Daxing District (Other); Tianjin Huanhu Hospital (Other); Guizhou Provincial People's Hospital (Other); Shandong Provincial Hospital (Other Government); The First Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Jining First People's Hospital (Other); Linyi People's Hospital (Other); Nanyang Central Hospital (Other); Rizhao People's Hospital (Other); Zhumadian Central Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Affiliated Hospital of Nantong University (Other); The Second Hospital of Anhui Medical University (Other); Changsha Central Hospital (Other); Jiujiang University Affiliated Hospital (Other Government); Liaocheng People's Hospital (Other); Chengde Central Hospital (Other Government); The First Affiliated Hospital of Anhui Medical University (Other); Jiangxi Provincial People's Hopital (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPENS-3
Record Dates: First submitted 2023-06-07; First posted 2023-07-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO group (Experimental): Normobaric Hyperoxia combined with intravenous thrombolysis
  Interventions: Procedure: Normobaric Hyperoxia; Drug: Intravenous thrombolysis(rt-PA)
- Control group (Placebo Comparator): Nasal oxygen combined with intravenous thrombolysis
  Interventions: Procedure: Nasal oxygen; Drug: Intravenous thrombolysis(rt-PA)

INTERVENTIONS:
Procedure: Normobaric Hyperoxia — Within 4.5 hours after stroke onset, patients were randomized into the NBO group and immediately given 100% oxygen inhalation (no more than 30 minutes after randomization) at a ventilation rate of 10L/ min using a sealed non-ventilating oxygen storage mask and keep giving oxygen for 4 hours. If the patient needs to be intubated with a ventilator to maintain ventilation, the FiO2 should be set to 1.0.
  Arms: NBO group
Procedure: Nasal oxygen — For nasal oxygen group, patients were immediately given oxygen inhalation (no more than 30 minutes after randomization) at a ventilation rate of 1L/min using nasal cannula and keep giving oxygen for 4 hours. If the patient needs to be intubated with a ventilator to maintain, the FiO2 should be set to 0.3 and gradualy incerased if spO2≤94%.
  Arms: Control group
Drug: Intravenous thrombolysis(rt-PA) — 10% dose of rt-PA (0.9 mg/kg) is given as bolus and the rest given as an infusion over the remaining 1 hour. Maximum dose 90mg.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Normobaric Hyperoxia combined with intravenous thrombolysis for acute ischemic stroke.

DETAILED DESCRIPTION:
In this study, cases of acute ischemic stroke who undergo intravenous thrombolysis within 4.5 hours from onset are included. The Normobaric Hyperoxia(NBO) group receive basic intravenous thrombolysis and given 100% oxygen inhalation at a ventilation rate of 10L/ min using a sealed non-ventilating oxygen storage mask and keep giving oxygen for 4 hours. The control group receive basic intravenous thrombolysis and given oxygen inhalation at a ventilation rate of 1L/min using nasal cannula and keep giving oxygen for 4 hours. The investigators aimed to determine the efficacy and safety of Normobaric Hyperoxia combined with intravenous thrombolysis for acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years;
2. The time from onset to randomization is within 4.5 hours of onset;
3. The clinical diagnosis is acute ischemic stroke (the criteria followed the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018);
4. Baseline NIHSS (at the time of randomization) should be ≥5 and ≤25 points;
5. Pre-stroke mRS score≤1 points;
6. Informed consent from the patient or surrogate.

Exclusion Criteria:

1. Intracranial hemorrhage (including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/extradural hematoma, etc.);
2. Past history of intracranial hemorrhage;
3. Rapid neurological function improvement, NIHSS score less than 5 points;
4. Presence of proximal arterial occlusion on computed tomographic angiography(CTA)/magnetic resonance angiography(MRA) (e.g., intracranial internal carotid artery(ICA), middle cerebral artery(MCA)-M1, and vertebrobasilar arteries);
5. Massive anterior cerebral infarction identified by CT or MRI (ASPECT < 6 or lesions larger than one third of the territory of the middle cerebral artery);
6. Intended to proceed endovascular treatment;
7. Pregnant women, or planning to become pregnant during the trial;
8. A history of severe head trauma or stroke within 3 months;
9. A history of intracranial or spinal surgery within 3 months;
10. A history of gastrointestinal or urinary bleeding within 3 weeks;
11. two weeks of major surgery;
12. Arterial puncture was performed at the hemostasis site that was not easily compressed within 1 week;
13. Active visceral bleeding;
14. Intracranial tumors, large intracranial aneurysms;
15. Aortic arch dissection was found;
16. Severe, sustained hypertension (Systolic Blood Pressure >185 mmHg or Diastolic Blood Pressure >110 mmHg);
17. Baseline blood glucose of <50mg/dL (2.78 mmol) or >400mg/dL (22.20 mmol);
18. Oral warfarin anticoagulant with international normalized ratio(INR)>1.7 or prothrombin time(PT)>15 s;
19. Heparin treatment was received within 24 h;
20. Thrombin inhibitors or factor Xa inhibitors were used within 48 h;
21. Propensity for acute bleeding, including platelet counts of less than 100×109/ L or otherwise;
22. Hereditary or acquired bleeding constitution;
23. Onset with seizures;
24. Severe liver and kidney dysfunction;
25. Active and chronic obstructive pulmonary disease or acute respiratory distress syndrome;
26. Patients with anemia or polycythemia vera or other situations that require urgent oxygen inhalation;
27. Patients with upper gastrointestinal bleeding or nausea or vomiting so that they cannot cooperate with the mask to inhale oxygen;
28. Life expectancy < 1 year;
29. Patients who could not complete the 90-day follow-up;
30. Participation in other clinical trials within 3 months prior to screening;
31. Unsuitability or participation in this study as judged by the Investigator may result in subjects being exposed to greater risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1230 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Utility-weighted modified Rankin scale scores | 90±7 days after randomization
  Utility-weighted modified Rankin scale scores

SECONDARY OUTCOMES:
Cerebral infarct volume | 24-48hours after randomization
  The infarct volume of cerebral infarct is evaluated by MRI
modified rankin scale (mRS) score | 90±7 days after randomization
  Ordinal distribution of mRS at 90±7 days after randomization;mRS score ranges from 0 to 5, and the higher score means a worse outcome
Good functional outcome | 90 ± 7 days after randomization
  Proportion of subjects with modified rankin scale (mRS) 0-2 at 90±7 days after randomization;mRS score ranges from 0 to 5, and the higher score means a worse outcome
Proportion of subjects with modified rankin scale (mRS) 0-3 | 90 ± 7 days after randomization
  Proportion of subjects with mRS 0-3 at 90±7 days after randomization;mRS score ranges from 0 to 5, and the higher score means a worse outcome
Scores assessed by National Institutes of Health Stroke Scale(NIHSS) | 4 ± 2 hours, 24 ± 6 hours, 72 ± 24 hours, 7 ± 2 days after randomization
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits
The proportion of neurological function improvement | 24 ± 6 hours after randomization
  ≥ 4 point reduction in National Institutes of Health Stroke Scale (NIHSS) score from baseline at 24 ± 6 hours after randomization;NIHSS score ranges from 0 to 42, and higher scores mean a worse outcome
Proportion of subjects with modified rankin scale (mRS) 0-1 | 30 ± 7 days after randomization
  Proportion of subjects with mRS 0-1 at 30±7 days after randomization;mRS score ranges from 0 to 5, and the higher score means a worse outcome
Barthel Index (BI) | 30 ± 7 days,90 ± 7 days after randomization
  The BI is an ordinal disability score of 10 categories (range from 0 to 100, higher values indicate better prognosis)
EuroQol five dimensions questionnaire（EQ-5D） | baseline before randomization,7 ± 2 days,30 ± 7 days,90 ± 7 days after randomization
  The score ranges from 0 to 100, with higher scores indicating optimal health
Days of hospitalization | 30 ± 7 days after randomization
  Length of stay in hospital
Stroke-related mortality | 90 ± 7 days after randomization
  Safety endpoint; the proportion of stroke related deaths in each group
All-cause mortality | 90 ± 7 days after randomization
  Safety endpoint; the proportion of all patients who died in each group
Symptomatic intracranial hemorrhage | 24 ± 6 hours after randomization
  Proportion of subjects with symptomatic intracranial hemorrhage at 24 ± 6 hours after randomization (defined by ECASSII and ECASS III)
Asymptomatic intracranial hemorrhage | 24 ± 6 hours after randomization
  The incidence of asymptomatic intracranial hemorrhage at 24 ± 6 hours after randomization
PH2 intracranial hemorrhage | 24 ± 6 hours after randomization
  The incidence of PH2 intracranial hemorrhage at 24 ± 6 hours after randomization (according to SITS standards)
Any intracranial hemorrhage | 24 ± 6 hours after randomization
  The incidence of any intracranial hemorrhage at 24 ± 6 hours after randomization
Systematic bleeding | 24 ± 6 hours after randomization
  The incidence of systematic bleeding at 24 ± 6 hours after randomization
Early neurological deterioration | 24 ± 6 hours after randomization
  Safety endpoint; defined as ≥4 point increase in National Institutes of Health Stroke Scale (NIHSS) score from baseline;NIHSS score ranges from 0 to 42, and higher scores mean a worse outcome
Oxygen-related adverse events | 90 ± 7 days after randomization
  Safety endpoint; the proportion of oxygen-related adverse events in each group, including severe lung infection, pneumothorax, atelectasis, respiratory failure, acute respiratory distress syndrome, and cardiopulmonary arrest
Adverse events/serious adverse events | 24 ± 12 hours, 7 ± 2 days, 90± 7 days after randomization
  Safety endpoint; the proportion of adverse events/serious adverse events in each group
PaO2 of arterial blood gas analysis | after 4 hours of oxygen therapy
  Safety endpoint
PaCO2 of arterial blood gas analysis | after 4 hours of oxygen therapy
  Safety endpoint
Potential of hydrogen(PH) of arterial blood gas analysis | after 4 hours of oxygen therapy
  Safety endpoint
Concentration of Lactic acid of arterial blood gas analysis | after 4 hours of oxygen therapy
  Safety endpoint
Systolic and diastolic blood pressure | 24 ± 6 hours after randomization
  Safety endpoint; vital signs
Heart rate | 24 ± 6 hours after randomization
  Safety endpoint; vital signs
Respiratory rate | 24 ± 6 hours after randomization
  Safety endpoint; vital signs
Oxygen saturation | 24 ± 6 hours after randomization
  Safety endpoint; vital signs
Unit costs | 7 ± 2 days, 30 ± 7 days,90 ± 7 days after randomization
  Unit costs will be attached to resource use, patient-reported and from hospital records after randomization, to obtain a cost per patient over the period of follow-up
Excellent functional outcome | 90±7 days after randomization
  Proportion of subjects with modified Rankin Scale(mRS) 0-1 at 90±7 days after randomization;mRS score ranges from 0 to 5, and the higher score means a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Xuan Wu Hospital，Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No